CLINICAL TRIAL: NCT03244137
Title: Effects of Pulmonary Rehabilitation on Cognitive Function in Patients With Severe to Very Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Collaborators: CHU de Rouen - Accueil (Other); Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: PR-COPD
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary rehabilitation: The whole population will benefit from a comprehensive pulmonary rehabilitation program, including aerobic training, superior and inferior limb strength training, self-management and add-on to pulmonary rehabilitation as needed (i.e : electrical muscle stimulation, inspiratory muscle training, non-invasive ventilation, high flow nasal canula).
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — See group description.

SUMMARY:
Chronic obstructive pulmonary disease is a leading cause of mortality worldwide.

It is a systemic disease which includes pulmonary, cardiac, muscular, digestive and cognitive impairments.

Pulmonary rehabilitation is a symptomatic treatment to reduce dyspnea and functional incapacity. However, it effects on cognitive dysfunction are not well known.

The aim of this study is to assess the effects of a comprehensive pulmonary rehabilitation program on cognitive dysfunction in patients with severe to very severe chronic obstructive pulmonary disease using the Montreal Cognitive Assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years;
* Chronic obstructive pulmonary disease stade III to IV;
* Referred for pulmonary rehabilitation.

Non Inclusion Criteria:

* Pregnancy or likely to be;
* History of psychiatric, neuro-vascular, cognitive disease or cranial trauma;
* Active alcoholism;
* Guardianship;
* Hospitalisation for acute exacerbation of chronic obstructive pulmonary disease in the previous 4 weeks;

Exclusion Criteria:

* Interruption of the pulmonary rehabilitation program > 15 days;
* Disruption of the training before the 18th session;
* Less than 18 sessions in four month.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Every patients with chronic obstructive pulmonary disease referred for pulmonary rehabilitation in ADIR Association (Rouen, France) and the Groupe Hospitalier du Havre (Le Havre, France) will be assessed for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Baseline cognitive function | Cognitive function is assessed at the beginning of the rehabilitation program : day 0
  Cognitive function is assessed with the Montreal Cognitive Assessement tool
Cognitive function after pulmonary rehabilitation | Cognitive function is assessed at the end of the rehabilitation program : day 60
  Cognitive function is assessed with the Montreal Cognitive Assessement tool
Cognitive function : follow up | Cognitive function is assessed 3 month after rehabilitation : day 150
  Cognitive function is assessed with the Montreal Cognitive Assessement tool
Change in cognitive function from baseline to the end of pulmonary rehabilitation | Change in cognitive function from baseline to the end of pulmonary rehabilitation is assessed with end of pulmonary rehabilitation minus baseline values (day 60 - day 0)
  Cognitive function is assessed with the Montreal Cognitive Assessement tool
Change in cognitive function from the end of pulmonary rehabilitation to 3 month of follow up | Change in cognitive function from the end of pulmonary rehabilitation to 3 month of follow up is assessed with the 3 month of follow minus the end of pulmonary rehabilitation values (day 150 - day 60)
  Cognitive function is assessed with the Montreal Cognitive Assessement tool

SECONDARY OUTCOMES:
Anxiety and depression : baseline | Anxiety and depression are assessed at the beginning of the rehabilitation program : day 0
  Anxiety and depression are assessed with the Hospital Anxiety and Depression scale (HAD).
Anxiety and depression : end of pulmonary rehabilitation | Anxiety and depression are assessed at the end of the rehabilitation program : day 60
  Anxiety and depression are assessed with the Hospital Anxiety and Depression scale (HAD).
Anxiety and depression : follow up | Anxiety and depression are assesses 3 month after the end of pulmonary rehabilitation program : day 150
  Anxiety and depression are assessed with the Hospital Anxiety and Depression scale (HAD).
Quality of life : baseline | Quality of life is assessed at the beginning of the rehabilitation program : day 0
  Quality of life is assessed using the Saint Georges Respiratory Questionnaire
Quality of life : end of pulmonary rehabilitation | Quality of life is assessed at the end of the rehabilitation program : day 60
  Quality of life is assessed using the Saint Georges Respiratory Questionnaire
Quality of life : follow-up | Quality of life is assessed 3 month after the end of the rehabilitation program : day 150
  Quality of life is assessed using the Saint Georges Respiratory Questionnaire
Functional capacity (six-minute stepper test) : baseline | Functional capacity is assessed at the beginning of the rehabilitation program : day 0
  Functional capacity is assessed with the six-minute stepper test
Functional capacity (six-minute stepper test) : end of pulmonary rehabilitation | Functional capacity is assessed at the end of the rehabilitation program : day 60
  Functional capacity is assessed with the six-minute stepper test
Functional capacity (six-minute walk test) : baseline | Functional capacity is assessed at the beginning of the rehabilitation program : day 0
  Functional capacity is assessed with the six-minute walk test
Adherence | Adherence is assessed at the end of the rehabilitation program : day 60
  Adherence to the pulmonary rehabilitation program is assessed by the following equation : number of session performed divided by the number of scheduled sessions
Relation between the cognitive function and the respiratory function (forced expiratory volume in 1 second) | The relation is assessed between baseline demographic data at day 0
  Cognitive function is assessed with the Montreal Cognitive Assessement tool and respiratory function is assessed with spirometric evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Cuvelier Antoine, Prof, PhD, Principal Investigator — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.; Muir Jean-François, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France.; Tardif Catherine, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Viacroze Catherine, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; Debeaumont David, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France.; Patout Maxime, MD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; Lamia Bouchra, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France.; Quieffin Jean, MD, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers.; Prieur Guillaume, PT, MsC, Study Chair — Service de pneumologie, Groupe Hospitalier du Havre, Fr; Médrinal Clément, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France; Gravier Francis-Edouard, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Bonnevie Tristan, PT, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.
Locations (2):
- France (2):
  - Bonnevie, Bois-Guillaume
  - Médrinal, Le Havre